CLINICAL TRIAL: NCT06237296
Title: A Phase I, Dose-escalation, Parallel-group, Randomized, Multi-center Study to Assess Safety and Immunogenicity of an RSV/hMPV mRNA Vaccine Candidate in Healthy Participants Aged 18 to 49 Years and 60 Years and Older.
Brief Title: Study of the Safety and Immune Response of an Investigational mRNA Vaccine for the Prevention of Respiratory Syncytial Virus and/or Human Metapneumovirus in Participants Aged 18 to 49 Years and 60 Years and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAV00027; VAV00027 (Other: Sanofi Identifier); U1111-1295-2931 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Syncytial Virus Infection; Healthy Volunteers; Metapneumovirus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: * Participants, Investigators and site staff remain blinded during study conduct, except dedicated study staff preparing/administering the study intervention.
  * Sponsor study staff will remain unblinded, except laboratory staff who handle primary/secondary endpoints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- RSV/hMPV mRNA / LNP 1 Group 1 (Experimental): Participants will be randomized to receive a single IM injection of RSV/hMPV mRNA / LNP vaccine 1 dose 1.
  Interventions: Biological: RSV/hMPV mRNA LNP 1
- RSV/hMPV mRNA / LNP 1 Group 2 (Experimental): Participants will be randomized to receive a single IM injection of RSV/hMPV mRNA / LNP vaccine 1 dose 2.
  Interventions: Biological: RSV/hMPV mRNA LNP 1
- RSV/hMPV mRNA / LNP 1 Group 3 (Experimental): Participants will be randomized to receive a single IM injection of RSV/hMPV mRNA / LNP vaccine 1 dose 3.
  Interventions: Biological: RSV/hMPV mRNA LNP 1
- RSV/hMPV mRNA / LNP 2 Group 4 (Experimental): Participants will be randomized to receive a single IM injection of RSV/hMPV mRNA / LNP vaccine 2 dose 1.
  Interventions: Biological: RSV/hMPV mRNA LNP 2
- RSV mRNA / LNP 1 Group 5 (Experimental): Participants will be randomized to receive a single IM injection of RSV mRNA / LNP vaccine 1 dose 1.
  Interventions: Biological: RSV mRNA LNP 1
- hMPV mRNA / LNP 1 Group 6 (Experimental): Participants will be randomized to receive a single IM injection of hMPV mRNA / LNP vaccine 1 dose 1.
  Interventions: Biological: hMPV mRNA LNP 1
- RSV/hMPV mRNA / LNP 1 Group 7 (Experimental): Participants will be randomized to receive a single IM injection of RSV/hMPV mRNA / LNP vaccine 1 dose 4.
  Interventions: Biological: RSV/hMPV mRNA LNP 1

INTERVENTIONS:
Biological: RSV/hMPV mRNA LNP 1 — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular Injection
  Arms: RSV/hMPV mRNA / LNP 1 Group 1; RSV/hMPV mRNA / LNP 1 Group 2; RSV/hMPV mRNA / LNP 1 Group 3; RSV/hMPV mRNA / LNP 1 Group 7
Biological: RSV/hMPV mRNA LNP 2 — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular Injection
  Arms: RSV/hMPV mRNA / LNP 2 Group 4
Biological: RSV mRNA LNP 1 — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular Injection
  Arms: RSV mRNA / LNP 1 Group 5
Biological: hMPV mRNA LNP 1 — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular Injection
  Arms: hMPV mRNA / LNP 1 Group 6

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity an investigational messenger ribonucleic acid (mRN)A vaccine for the prevention of lower respiratory tract disease (LRTD) caused by respiratory syncytial virus (RSV) and/or human metapneumovirus (hMPV) in older adults. A single intramuscular (IM) injection of 3 to 4 different doses of the RSV/hMPV mRNA vaccine candidate formulated with 2 different lipid nanoparticles (LNP) will be administered to healthy participants aged 18 to 49 years and 60 years and older.

Treatment:

* RSV/hMPV mRNA / LNP 1 at 3-4 different doses or,
* RSV/hMPV mRNA / LNP 2 at 3-4 difference doses or,
* RSV mRNA / LNP 1 at 1 dose or,
* hMPV mRNA / LNP 1 at 1 dose

DETAILED DESCRIPTION:
Study duration per participant is approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

-Informed consent form (ICF) has been signed and dated

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

-Any condition which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

--The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Presence of unsolicited systemic immediate adverse events (AEs) | Within 30 minutes after vaccination
  Number of participants experiencing immediate an immediate unsolicited systemic adverse event
Presence of solicited injection site or systemic reactions | Within 7 days after vaccination
  Number of participants reporting:
  * injection site reactions: pain, erythema and swelling
  * systemic reactions: fever, headache, fatigue, myalgia, arthralgia and chills
Presence of unsolicited AEs | Within 28 days after vaccination
  Number of participants experiencing unsolicited AEs
Presence of medically attended adverse events (MAAEs) | Throughout study (up to approximately 6 months)
  Number of participants experiencing MAAEs
Presence of serious adverse events (SAEs) | Throughout study (up to approximately 6 months)
  Throughout study (up to approximately 6 months)
Presence of adverse events of special interest (AESIs) | Throughout study (up to approximately 6 months)
  Number of participants experiencing AESIs
Presence of out-of-range biological test results | Within 7 days after vaccination
  Number of participants with biological safety assessment values out of normal range (as per the laboratory performing the test, including shift from baseline values)
RSV-A serum neutralizing antibody (nAb) titers at pre-vaccination (D01) and 28 days post- vaccination (D29) in the RSV/hMPV and monovalent RSV formulations | Day 1 and Day 29
  RSV-A serum nAb titers at pre-vaccination (D01), 28 days (D29) post-vaccination
RSV-B serum neutralizing antibody (nAb) titers at pre-vaccination (D01) and 28 days post- vaccination (D29) in the RSV/hMPV and monovalent RSV formulations | Day 1 and Day 29
  RSV-B serum nAb titers at pre-vaccination (D01), 28 days (D29) post-vaccination
hMPV- A serum neutralizing antibody (nAb) titers at pre-vaccination (D01) and 28 days post- vaccination (D29) in the RSV/hMPV and monovalent hMPV formulations | Day 1 and Day 29
  hMPV-A serum nAb titers at pre-vaccination (D01), 28 days (D29) post-vaccination

SECONDARY OUTCOMES:
RSV A serum nAb titers at pre vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination in the monovalent RSV formulation | Day 1, Day 29, Day 91 and Day 181
  RSV A serum nAb titers at pre vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination
RSV B serum nAb titers at pre vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination in the monovalent RSV formulation | Day 1, Day 29, Day 91 and Day 181
  RSV B serum nAb titers at pre vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination
RSV A serum anti-F immunoglobulin G (IgG) antibody (Ab) titers at pre-vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination in the monovalent RSV formulation | Day 1, Day 29, Day 91 and Day 181
  RSV A serum anti-F immunoglobulin G (IgG) antibody (Ab) titers at pre-vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination
hMPV A serum nAb titers at pre vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination in the monovalent hMPV formulations | Day 1, Day 29, Day 91 and Day 181
  hMPV A serum nAb titers at pre vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination
hMPV A serum anti-F IgG Ab titers at pre vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination in the monovalent hMPV formulations | Day 1, Day 29, Day 91 and Day 181
  hMPV A serum anti-F IgG Ab titers at pre vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - Velocity Gardena Site Number : 8400011, Gardena, California
  - Velocity Clinical Research-Hallandale Beach- Site Number : 8400013, Hallandale, Florida
  - Advanced Clinical Research- Site Number : 8400005, Meridian, Idaho
  - Velocity Clinical Research, Sioux City Site Number : 8400017, Sioux City, Iowa
  - Velocity Clinical Research- New Orleans Site Number : 8400016, New Orleans, Louisiana
  - Meridian Clinical Research- Site Number : 8400007, Binghamton, New York
  - Velocity Clinical Research- Site Number : 8400012, Cleveland, Ohio
  - Coastal Carolina Research Center- Site Number : 8400001, North Charleston, South Carolina
  - Charlottesville Medical Research Center Winding River - Site Number : 8400002, Charlottesville, Virginia
- Australia (8):
  - Investigational Site Number : 0360006, Blacktown, New South Wales
  - Investigational Site Number : 0360002, Botany, New South Wales
  - Investigational Site Number : 0360003, Kanwal, New South Wales
  - Investigational Site Number : 0360004, Sydney, New South Wales
  - Investigational Site Number : 0360008, Herston, Queensland
  - Investigational Site Number : 0360005, Morayfield, Queensland
  - Investigational Site Number : 0360001, Camberwell, Victoria
  - Investigational Site Number : 0360007, Canberra

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAV00027 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25593&tenant=MT_SNY_9011